CLINICAL TRIAL: NCT00157209
Title: A Multicenter Phase IIb Randomised, Controlled Study of BLP25 Liposome Vaccine for Active Specific Immunotherapy of Non-Small Cell Lung Cancer
Brief Title: Phase 2b Randomized Controlled Study of Tecemotide (L-BLP25) for Immunotherapy of NSCLC (Non-Small Cell Lung Cancer)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B25-LG-304 / EMR 63325-005
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Lung Neoplasms; Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — L-BLP25; Single Person; Cyclophosphamide

ARMS (2):
- Tecemotide (L-BLP25) plus Best Supportive Care (BSC) (Experimental)
  Interventions: Biological: Tecemotide (L-BLP25); Drug: Single low dose cyclophosphamide; Other: Best Supportive Care (BSC)
- Best Supportive Care (BSC) Alone (Active Comparator)
  Interventions: Other: Best Supportive Care (BSC)

INTERVENTIONS:
Biological: Tecemotide (L-BLP25) — After receiving single low dose cyclophosphamide, subjects will receive 8 consecutive weekly subcutaneous vaccinations with 1000 microgram (mcg) of tecemotide (L-BLP25) at weeks 0, 1, 2, 3, 4, 5, 6 and 7 followed by maintenance vaccinations (1000 mcg of tecemotide (L-BLP25) at 6-week intervals, commencing at Week 13, until discontinuation from the study due to ECOG status of 4, participation in alternate trial, serious adverse event, or reasons that preclude assessment of clinical status in the opinion of the investigator, and in case of unavailability of study vaccine.
  Arms: Tecemotide (L-BLP25) plus Best Supportive Care (BSC)
Drug: Single low dose cyclophosphamide — A single intravenous infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide will be given 3 days before the first vaccine treatment.
  Arms: Tecemotide (L-BLP25) plus Best Supportive Care (BSC)
Other: Best Supportive Care (BSC) — The BSC will be provided at the investigator's discretion, and may include palliative radiation, psychosocial support, analgesics and nutritional support. Second-line chemotherapy is permitted when indicated for treatment of progressive disease.

SUMMARY:
This is a prospective open label, controlled, randomized study to test the safety and efficacy of active specific immunotherapy with tecemotide (L-BLP25) for the treatment of subjects with Stage IIIB or Stage IV non-small cell lung cancer (NSCLC). To be eligible, subjects entering the trial will have to demonstrate either stable disease or a clinical response after first-line treatment (chemotherapy alone, or chemotherapy and radiotherapy) and have an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2. Following a 3 week washout period, subjects will be stratified by disease status (either Stage IIIB locoregional disease or Stage IIIB with malignant pleural effusion and Stage IV), and randomized to either best supportive care (BSC) plus tecemotide (L-BLP25) treatment or BSC alone.

ELIGIBILITY:
Inclusion Criteria:

* Stage IIIB or Stage IV NSCLC
* Stable disease or a clinical response following first-line treatment, consisting of either chemotherapy alone or chemotherapy and radiotherapy. Subjects must have completed the first-line treatment at least 3 weeks prior to study entry
* Eastern Cooperative Oncology Group (ECOG) performance status of greater than or equal to (>=) 2
* Ability to understand and willingness to sign a written informed consent
* Other protocol-defined inclusion criteria could apply

Exclusion Criteria:

* Received immunotherapy within 4 weeks prior to study entry
* Received immunosuppressive drugs within 3 weeks prior to study entry
* Subjects with known brain metastases
* Past or current history of neoplasm other than lung carcinoma, except for curatively treated non-melanoma skin cancer, in situ carcinoma of the cervix or other cancer curatively treated and with no evidence of disease for at least 5 years
* Autoimmune disease or immunodeficiency
* Clinically significant hepatic, renal or cardiac dysfunction
* Subjects with clinically significant active infection
* Pregnant or breast feeding women, women of childbearing potential, unless using effective contraception as determined by the investigator
* Other protocol-defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2000-08; Primary Completion 2006-03 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Please Contact the Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- [Result] Butts C, Murray N, Maksymiuk A, Goss G, Marshall E, Soulieres D, Cormier Y, Ellis P, Price A, Sawhney R, Davis M, Mansi J, Smith C, Vergidis D, Ellis P, MacNeil M, Palmer M. Randomized phase IIB trial of BLP25 liposome vaccine in stage IIIB and IV non-small-cell lung cancer. J Clin Oncol. 2005 Sep 20;23(27):6674-81. doi: 10.1200/JCO.2005.13.011. PMID 16170175
- [Result] Butts C, Maksymiuk A, Goss G, Soulieres D, Marshall E, Cormier Y, Ellis PM, Price A, Sawhney R, Beier F, Falk M, Murray N. Updated survival analysis in patients with stage IIIB or IV non-small-cell lung cancer receiving BLP25 liposome vaccine (L-BLP25): phase IIB randomized, multicenter, open-label trial. J Cancer Res Clin Oncol. 2011 Sep;137(9):1337-42. doi: 10.1007/s00432-011-1003-3. Epub 2011 Jul 9. PMID 21744082
- [Result] Butts C, Maksymiuk A, Goss G, et al. A multi-centre phase IIB randomized controlled study of BLP25 liposome vaccine (L-BLP25 or Stimuvax) for active specific immunotherapy of non-small cell lung cancer (NSCLC): updated survival analysis. J Thoracic Oncol. 2007 Aug; 2(8), Suppl 4, S332-3.
- [Result] Butts C, Anderson H, Maksymiuk A, et al. Long-term safety of BLP25 liposome vaccine (L-BLP25) in patients (pts) with stage IIIB/IV non-small cell lung cancer (NSCLC). J Clin Onc 2009; 27(15S): abstract 3055.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First/Last participant (informed consent): 08 August 2000/02 December 2002. Clinical data cut-off: 15 March 2006. Participants randomized at 17 centers in Canada and United Kingdom.
Pre-assignment Details: A total of 437 participants were screened for eligibility and 171 participants were randomized.
Groups:
- Tecemotide (L-BLP25) Plus Best Supportive Care (BSC): A single intravenous infusion of 300 milligram per square meter (mg/m^2) (to a maximum 600 mg) of cyclophosphamide was given 3 days before the first vaccine treatment. After receiving cyclophosphamide, participants received 8 consecutive weekly subcutaneous vaccinations with 1000 microgram (mcg) of tecemotide (L-BLP25) at Weeks 0, 1, 2, 3, 4, 5, 6, and 7 followed by maintenance vaccinations with 1000 mcg of tecemotide (L-BLP25) at 6-week intervals, commencing at Week 13, until discontinuation from study due to ECOG status of 4, participation in alternate trial, serious adverse event, or reasons that preclude assessment of clinical status in the opinion of investigator, and incase of unavailability of study vaccine. The Best Supportive Care (BSC) was provided at the investigator's discretion, and included palliative radiation, psychosocial support, analgesics and nutritional support as required. Second-line chemotherapy was permitted when indicated for treatment of progressive disease.
- Best Supportive Care (BSC) Alone: The BSC was provided at the investigator's discretion, and included palliative radiation, psychosocial support, analgesics and nutritional support as required. Second-line chemotherapy was permitted when indicated for treatment of progressive disease.
Period: Overall Study
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone
Started | 88 | 83
Completed | 78 | 83
Not Completed | 10 | 0
Not completed — Ongoing at data cut-off | 10 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone | Total
Number analyzed (Participants) | 88 | 83 | 171
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (10.0) | 58.7 (11.3) | 59.6 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 40 | 76
  Male | 52 | 43 | 95

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, and TEAEs With Cancer and Leukemia Group B (CALGB) Toxicity Grade 3 or 4
Description: An adverse event (AE) was defined as any new untoward medical occurrences/worsening of pre-existing medical condition, whether or not related to study drug. A serious AE was an AE that results in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect. Treatment-emergent are events between first dose of study drug and up to 30 days after last dose that were absent before treatment or that worsened relative to pretreatment state. Number of participants with TEAEs, serious TEAEs, TEAEs leading to death, and TEAEs with CALGB toxicity Grade 3 or 4 were reported.
Time Frame: From the first dose of study drug administration until 30 days after the last dose of study drug administration or assessed until cut-off date (15 March 2006)
Population: Analysis population included all participants randomized in the study.
Measure: Number; unit: participants
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone
Number analyzed (Participants) | 88 | 83
participants
  TEAEs | 88 | 80
  Serious TEAEs | 29 | 34
  TEAEs leading to death | 13 | 20
  TEAEs with CALGB toxicity Grade 3 or 4 | 42 | 42

2. Primary Outcome: Overall Survival Time
Description: Time from randomization to death or last day known to be alive. Participants without event were censored at the last date known to be alive or at the clinical cut-off date (15 March 2006), whichever was earlier.
Time Frame: Time from randomization to death or last day known to be alive, reported between day of first participant randomized that is, 08 August 2000, up to cut-off (15 March 2006)
Population: Analysis population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone
Number analyzed (Participants) | 88 | 83
months | 17.2 [12.9 to 24.2] | 13.0 [11.2 to 16.2]
Statistical Analysis 1: Comparison: Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) vs Best Supportive Care (BSC) Alone; Test type: Superiority or Other; p = 0.045, Log Rank; Hazard Ratio (HR) = 0.745, 95% CI 2-sided [0.533 to 1.042]

3. Secondary Outcome: Functional Assessment of Cancer Therapy (FACT-L) Questionnaire Score
Description: Functional Assessment of Cancer Therapy - Lung cancer (FACT-L) is a valid instrument used to measure quality of life (QoL) in participants with cancer consisting of the 27-item FACT-General (G) and 9-item lung cancer subscale (LCS). FACT-G is organized into subscales: physical well-being (PWB)-7 items; social/family well-being (SWB)-7 items; emotional well-being (EWB)-6 items; functional well-being (FWB)-7 items. Each item uses a 5 point rating scale (0="not at all" and 4=equals "very much"). FACT-L total score=4 subscales + LCS and ranges from 0 to 144. Higher scores indicate better QOL.
Time Frame: At baseline, Week 4, Week 8 and then at 12 Week intervals beginning at week 19 until withdrawal/discontinuation from the study.
Population: Analysis population included all the participants with a baseline and at least one post-baseline complete FACT-L questionnaire. "n" signifies number of participants evaluable at each timepoint for this outcome measure, for each reporting group, respectively.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone
Number analyzed (Participants) | 88 | 78
Units on a scale
  Baseline (n=88, 78) | 109.3 (14.8) | 106.4 (15.6)
  Week 4 (n=86, 75) | 109.4 (15.9) | 104.1 (17.0)
  Week 8 (n=84, 73) | 108.1 (16.1) | 101.6 (17.5)
  Week 19 (n=54, 55) | 108.2 (14.9) | 100.1 (20.6)
  Week 31(n=34, 36) | 110.1 (14.7) | 103.5 (19.6)
  Week 43 (n=31, 20) | 110.3 (17.4) | 111.6 (12.8)

4. Secondary Outcome: Number of Participants With Positive T-cell Proliferation
Description: T-cell proliferation assays were performed and the number of participants with positive mucinous glycoprotein 1 (MUC1) specific T-cell proliferative response were reported.
Time Frame: Time from randomization until cut-off date (15 March 2006)
Population: Analysis population included all randomized participants. "N" signifies total number of participants who were evaluable for this measure. T-cell measure was done only on arm A where subjects received tecemotide for induction of t-cell response. Therefore arm B BSC did not have any samples taken for this assessment.
Measure: Number; unit: participants
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone
Number analyzed (Participants) | 78 | 0
participants | 16 |

5. Secondary Outcome: Number of Participants With Elevated CA27-29 Antigen Levels
Description: CA 27-29 is a blood test used to monitor certain types of cancer. CA 27-29 is the name of an antigen, which is a substance that stimulates your body's defense system. CA27-29 antigen levels were determined on all participants and assessed the disease burden of participants at study entry, evaluated early recurrence, presence of residual disease, continued remission or poor prognosis.
Time Frame: Study entry, Week 8
Population: Analysis population included all randomized participants. "n" signifies number of participants evaluable at each timepoint for this outcome measure, for each reporting group, respectively.
Measure: Number; unit: participants
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone
Number analyzed (Participants) | 88 | 83
participants
  Study entry (n=84, 82) | 21 | 21
  Week 8 (n=82, 71) | 20 | 18

ADVERSE EVENTS:
Time Frame: From the first dose of study drug administration until 30 days after the last dose of study drug administration or assessed until cut-off date (15 March 2006)
Description: A serious adverse event was an AE that resulted in any of the following outcomes: death, life threatening, persistent/significant disability/incapacity, initial or prolonged inpatient hospitalization, congenital anomaly/birth defect.
Arm/Group | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) | Best Supportive Care (BSC) Alone
Serious Adverse Events (participants affected / at risk) | 29/88 | 34/83
Other Adverse Events (participants affected / at risk) | 88/88 | 80/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) (N=88) | Best Supportive Care (BSC) Alone (N=83)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 6
Metastases to brain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer stage unspecified (excl metastatic tumours to lung) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung squamous cell carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm NOS, primary site unknown (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumothorax NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia NOS (Infections and infestations) | 2 | 3
Lower respiratory tract infection NOS (Infections and infestations) | 1 | 1
Bronchopneumonia NOS (Infections and infestations) | 0 | 1
Empyema NOS (Infections and infestations) | 1 | 0
Sepsis NOS (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 4
Cardiac arrest (Cardiac disorders) | 1 | 1
Myocardial infarction (Cardiac disorders) | 0 | 2
Angina unstable (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage NOS (Gastrointestinal disorders) | 0 | 2
Abdominal pain NOS (Gastrointestinal disorders) | 1 | 0
Intestinal perforation NOS (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1
Fractured pelvis NOS (Injury, poisoning and procedural complications) | 1 | 0
Radiation injury NOS (Injury, poisoning and procedural complications) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Convulsions NOS (Nervous system disorders) | 0 | 1
Intracranial haemorrhage NOS (Nervous system disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Deep venous thrombosis NOS (Vascular disorders) | 1 | 0
Superior vena caval obstruction (Vascular disorders) | 1 | 0
Weakness (General disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia NOS (Metabolism and nutrition disorders) | 0 | 1
Renal failure NOS (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tecemotide (L-BLP25) Plus Best Supportive Care (BSC) (N=88) | Best Supportive Care (BSC) Alone (N=83)
Anaemia NOS (Blood and lymphatic system disorders) | 5 | 6
Tachycardia NOS (Cardiac disorders) | 2 | 5
Abdominal pain NOS (Gastrointestinal disorders) | 9 | 8
Abdominal pain upper (Gastrointestinal disorders) | 7 | 3
Constipation (Gastrointestinal disorders) | 15 | 17
Diarrhoea NOS (Gastrointestinal disorders) | 13 | 8
Dyspepsia (Gastrointestinal disorders) | 11 | 9
Dysphagia (Gastrointestinal disorders) | 6 | 5
Nausea (Gastrointestinal disorders) | 44 | 31
Vomiting NOS (Gastrointestinal disorders) | 18 | 17
Chest discomfort (General disorders) | 7 | 3
Chest pain (General disorders) | 26 | 13
Chest tightness (General disorders) | 8 | 2
Fatigue (General disorders) | 39 | 32
Fatigue aggravated (General disorders) | 6 | 8
Influenza like illness (General disorders) | 10 | 3
Injection site bruising (General disorders) | 19 | 0
Injection site erythema (General disorders) | 22 | 0
Injection site pain (General disorders) | 21 | 0
Injection site swelling (General disorders) | 7 | 0
Lethargy (General disorders) | 5 | 4
Nodule (General disorders) | 14 | 0
Oedema peripheral (General disorders) | 8 | 7
Pyrexia (General disorders) | 13 | 10
Rigors (General disorders) | 7 | 4
Weakness (General disorders) | 10 | 12
Bronchitis NOS (Infections and infestations) | 6 | 2
Herpes simplex (Infections and infestations) | 6 | 1
Influenza (Infections and infestations) | 6 | 0
Lower respiratory tract infection NOS (Infections and infestations) | 4 | 10
Nasopharyngitis (Infections and infestations) | 19 | 13
Oral candidiasis (Infections and infestations) | 1 | 6
Pneumonia NOS (Infections and infestations) | 5 | 3
Upper respiratory tract infection NOS (Infections and infestations) | 11 | 6
Weight decreased (Investigations) | 11 | 11
Anorexia (Metabolism and nutrition disorders) | 30 | 25
Appetite decreased NOS (Metabolism and nutrition disorders) | 4 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 20
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Muscle cramps (Musculoskeletal and connective tissue disorders) | 9 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 8 | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 10
Pain in limb (Musculoskeletal and connective tissue disorders) | 9 | 7
Shoulder blade pain (Musculoskeletal and connective tissue disorders) | 5 | 1
Dizziness (Nervous system disorders) | 15 | 9
Dysgeusia (Nervous system disorders) | 6 | 2
Headache NOS (Nervous system disorders) | 21 | 21
Hypoaesthesia (Nervous system disorders) | 12 | 13
Paraesthesia (Nervous system disorders) | 6 | 5
Anxiety (Psychiatric disorders) | 5 | 8
Depression (Psychiatric disorders) | 2 | 5
Insomnia (Psychiatric disorders) | 14 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 41 | 24
Cough aggravated (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 26 | 26
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 12 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 17 | 12
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 4
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 18 | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 5 | 14
Rash NOS (Skin and subcutaneous tissue disorders) | 13 | 4
Sweating increased (Skin and subcutaneous tissue disorders) | 10 | 3
Hypotension NOS (Vascular disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
By signing this protocol, the investigator affirms to the Sponsor that information furnished by the Sponsor will be maintained in confidence, and such information will be divulged to the IRB/IEC under an appropriate understanding of confidentiality with such a committee. It is required that copies of all papers, abstracts, articles, etc. that contain study data are to be forward to the Sponsor for review 30 days prior to submission for publication.